CLINICAL TRIAL: NCT00007397
Title: Age, Risk Factors for CVD and Cognitive Functioning
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 958; R43HL065117 (NIH)
Record Dates: First submitted 2000-12-19; First posted 2000-12-19 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2005-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Neurologic Manifestations
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Neurologic Manifestations

SUMMARY:
To relate cardiovascular disease (CHD) risk factors to cognitive performance among middle-aged and elderly men and women over a 10 year longitudinal study period.

DETAILED DESCRIPTION:
BACKGROUND:

The Framingham Heart Study is a major epidemiological investigation of prospective relationships between risk factors for the development of cardiovascular disease (CVD risk factors) and CVD risk factor outcomes. The Framingham Study and other large, prospective studies have resulted in an extensive literature on the impact of CVD risk factors (including age) and CVD outcomes. Comparatively, there have been many fewer studies of the impact of CVD risk factors on cognitive functioning, and possibly no studies of the effect of objectively measured, competing risk factors on cognitive functioning.

DESIGN NARRATIVE:

Dr. Elias and colleagues used cardiovascular risk factor data from the Framingham Heart Study (N= 2,123) in a prospective design allowing them to relate CVD risk factors (including age and gender) to two outcome measures: (1) level of cognitive performance and (2) change in cognitive performance over a 10 year longitudinal study period. The overall goals were to determine the best multivariate combination of biological and psychosocial risk factors for the prediction of lowered cognitive ability in middle-aged and elderly men and women, and to evaluate the relative impact of age, gender, and other biological and psychosocial risk factors on cognitive functioning.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-02; Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merrill Elias — Boston University

REFERENCES:
- [Background] Elias MF, Elias PK, Sullivan LM, Wolf PA, D'Agostino RB. Lower cognitive function in the presence of obesity and hypertension: the Framingham heart study. Int J Obes Relat Metab Disord. 2003 Feb;27(2):260-8. doi: 10.1038/sj.ijo.802225. PMID 12587008
- [Background] Elias MF, Sullivan LM, D'Agostino RB, Elias PK, Beiser A, Au R, Seshadri S, DeCarli C, Wolf PA. Framingham stroke risk profile and lowered cognitive performance. Stroke. 2004 Feb;35(2):404-9. doi: 10.1161/01.STR.0000103141.82869.77. Epub 2004 Jan 15. PMID 14726556
- [Background] Elias PK, Elias MF, D'Agostino RB, Sullivan LM, Wolf PA. Serum cholesterol and cognitive performance in the Framingham Heart Study. Psychosom Med. 2005 Jan-Feb;67(1):24-30. doi: 10.1097/01.psy.0000151745.67285.c2. PMID 15673620